CLINICAL TRIAL: NCT06846255
Title: Comparison of Successful Treatment Outcomes of Dexamethasone Cyclophosphamide Pulse (DCP) Therapy and Dexamethasone Azathioprine Pulse (DAP) Therapy in Pemphigus Vulgaris Patients At a Tertiary Care Hospital, Karachi
Brief Title: Comparing DCP and DAP for Pemphigus Vulgaris
Acronym: DCP;DAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Principal Investigator, Zainab Javed, Principal Investigator, Jinnah Postgraduate Medical Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 53727
Record Dates: First submitted 2025-02-24; First posted 2025-02-26 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Pemphigus Vulgaris
MeSH Terms: conditions — Pemphigus

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone Cyclophosphamide Pulse therapy group (DCP group) (Active Comparator): Patients were randomly assigned to two groups. The DCP group received therapy consisting of monthly doses of 100 mg dexamethasone dissolved in 500 ml of 5% dextrose, administered intravenously over 2 hours on 3 consecutive days. On the second day, 500 mg of cyclophosphamide was added in infusion. Between treatment cycles, patients took 50 mg of cyclophosphamide orally each day. This treatment regimen continued for 6 months, and outcomes were assessed after 3 treatment cycles.
  Interventions: Drug: Dexamethasone Cyclophosphamide Pulse therapy
- Dexamethasone Azathioprine Pulse therapy group (DAP group) (Active Comparator): Patients were randomly assigned to two groups. The DAP group received therapy consisting of monthly doses of 100 mg dexamethasone dissolved in 500 ml of 5% dextrose, administered intravenously over 2 hours on 3 consecutive days. Cyclophosphamide is replaced by daily oral azathioprine. No bolus dose of azathioprine is given. This treatment regimen continued for 6 months, and outcomes were assessed after 3 treatment cycles.
  Interventions: Drug: Dexamethasone Azathioprine Pulse therapy

INTERVENTIONS:
Drug: Dexamethasone Cyclophosphamide Pulse therapy — 33 patients were enrolled in DCP group. They were given Dexamethasone Cyclophosphamide pulse therapy for 6 months and successful treatment outcome was assessed using Pemphigus Disease Area Index (PDAI) scores.
  Other Names: Injection Decadron, Cytoxan pulse therapy
  Arms: Dexamethasone Cyclophosphamide Pulse therapy group (DCP group)
Drug: Dexamethasone Azathioprine Pulse therapy — 33 patients were enrolled in DAP group. They were given Dexamethasone Azathioprine pulse therapy for 6 months and successful treatment outcome was assessed using Pemphigus Disease Area Index (PDAI) scores.
  Other Names: Injection Decadron , Tablet Imuran Pulse therapy
  Arms: Dexamethasone Azathioprine Pulse therapy group (DAP group)

SUMMARY:
What's the study about?

This study focused on comparing two different treatments for pemphigus vulgaris, a skin condition caused when body's immune system works against itself. The treatments were dexamethasone cyclophosphamide pulse (DCP) therapy and dexamethasone azathioprine pulse (DAP) therapy.

Why was this study done?

The goal of the study was to determine which treatment, DCP or DAP, was more effective in treating pemphigus vulgaris. Both treatments involve high-dose steroids combined with other medications, but they differ in the specific medications used.

How did they do the study?

Researchers conducted a randomized controlled trial, where patients were randomly assigned to receive either DCP or DAP therapy. They then followed these patients to see how well each treatment worked.

DETAILED DESCRIPTION:
Consenting patients presenting with pemphigus vulgaris visiting Outpatient Department of Dermatology, Jinnah Postgraduate Medical Centre, Karachi, were enrolled in this study who fulfilled the inclusion criteria. Permission from the institutional ethical review committee were taken prior to conduction of study. Brief history was taken about the duration of pemphigus vulgaris, demographic data (age, gender and residence status) and written informed consent in local language (Urdu) was taken from each patient. Patients were randomly allocated using sealed opaque envelop bearing A= Dexamethasone cyclophosphamide pulse (DCP) therapy and B= and dexamethasone azathioprine pulse (DAP) therapy. Patients in group A received monthly doses of 100 mg of dexamethasone dissolved in 500 ml of 5% dextrose by slow intravenous infusion over 2 h on 3 consecutive days along with 500 mg of cyclophosphamide in the infusion on day 2. In between the pulses, patients received 50 mg of oral cyclophosphamide daily. Patients in group B, cyclophosphamide bolus dose on day 2 omitted, and a daily dose of 50 mg of azathioprine will be given throughout the pulses. Patient's blood pressure, pulse rate, heart rate was monitored every 15 min during the period of infusion. Serum electrolytes and electrocardiography was repeated after completion of each pulse. The cycles was repeated at 28-day interval starting from day 1 of the previous cycle. Response to both treatment regimens was evaluated after 3 cycle and successful treatment outcome was labeled as per operational definition. The findings of quantitative variable (age, mean PDAI score in group A and B, and duration of pemphigus vulgaris) and qualitative variables (gender, residence status, smoking status, family monthly income, occupational status and successful treatment outcome) was entered in a form.

Data was analyzed on Statistical Package for the Social Sciences software Version 22.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Pemphigus Vulgaris for more than one month
* Either gender
* Pemphigus Disease Area Index (PDAI) ≥ 15 points
* Age 20-60 years

Exclusion Criteria:

* History of Hepatitis C, B, or HIV infection
* History of connective tissue disorders, malignancy, diabetes mellitus, hypo/hyperthyroidism
* Pregnant patients
* History of congestive cardiac failure, chronic liver disease, asthma, chronic obstructive pulmonary disease and stroke

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Pemphigus Disease Area Index (PDAI) | Baseline, 3 months & 6 months
  Successful treatment outcome is assessed with Pemphigus Disease Area Index (PDAI) score. Lower score means better outcome

OTHER OUTCOMES:
Dermatology Life Quality Index | baseline, 3 months, 6 months
  Life quality of patients enrolled was assessed during study using Dermatology Life Quality Index (DLQI). Higher score means negative impact on patient's quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Zainab Javed, MBBS, Principal Investigator — Jinnah Postgraduate Medical Centre; Rabia Ghafoor, MBBS, FCPS, Study Chair — Jinnah Postgraduate Medical Centre
Locations (1):
- Jinnah Postgraduate Medical Center, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chryssomallis F, Dimitriades A, Chaidemenos GC, Panagiotides D, Karakatsanis G. Steroid-pulse therapy in pemphigus vulgaris long term follow-up. Int J Dermatol. 1995 Jun;34(6):438-42. doi: 10.1111/j.1365-4362.1995.tb04450.x. PMID 7657447
- [Background] Fernandes NC, Menezes M. Pulse therapy in pemphigus: report of 11 cases. An Bras Dermatol. 2013 Jul-Aug;88(4):672-5. doi: 10.1590/abd1806-4841.20131840. PMID 24068153
- [Background] Hassan I, Sameem F, Masood QM, Majid I, Abdullah Z, Ahmad QM. Non Comparative Study on Various Pulse Regimens (DCP, DAP and DMP) in Pemphigus: Our Experience. Indian J Dermatol. 2014 Jan;59(1):30-4. doi: 10.4103/0019-5154.123487. PMID 24470657
- [Background] Mustafi S, Sinha R, Hore S, Sen S, Maity S, Ghosh P. Pulse therapy: Opening new vistas in treatment of pemphigus. J Family Med Prim Care. 2019 Mar;8(3):793-798. doi: 10.4103/jfmpc.jfmpc_114_19. PMID 31041203